CLINICAL TRIAL: NCT01380769
Title: A Randomized, Phase 2, Study to Assess the Safety and Activity of CRLX101, a Nanoparticle Formulation of Camptothecin, in Patients With Advanced Non-Small Cell Lung Cancer Who Have Failed One or Two Previous Regimens of Chemotherapy
Brief Title: A Phase 2 Study of CRLX101(NLG207) in Patients With Advanced Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NewLink Genetics Corporation (Industry)
Responsible Party: Sponsor
Organization: Lumos Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRLX-002
Record Dates: First submitted 2011-06-22; First posted 2011-06-27 (Estimated); Results first posted 2017-05-24 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — IT-101

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CRLX101 (Experimental)
  Interventions: Drug: CRLX101
- Best supportive care (Other)
  Interventions: Other: Best Supportive Care

INTERVENTIONS:
Drug: CRLX101 — CRLX101 is administered at 15mg/m2 IV every other week
  Other Names: NLG207
  Arms: CRLX101
Other: Best Supportive Care — best supportive care
  Arms: Best supportive care

SUMMARY:
The purpose of this study is to compare median overall survival of patients with advanced non-small cell lung cancer (NSCLC) treated with CRLX101 to patients treated with best supportive care (BSC).

DETAILED DESCRIPTION:
Lung cancer remains the leading cause of cancer-related mortality in men and women worldwide. Non-small cell lung cancer (NSCLC) accounts for approximately 80% of all lung cancer. The development of targeted therapies has changed the approach to treating NSCLC significantly over the past decade with targeted therapies generally possessing safety advantages over traditional cytotoxic regimens. However, combination paradigms and resistance patterns complicate the use of these agents. CRLX101 is a nanoparticle comprised of camptothecin (CPT) conjugated to a cyclodextrin-based polymer. CRLX101 is designed to increase the exposure of tumor cells to CPT while minimizing side effects.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients who are ≥ 18-years of age.
* Histologically or cytologically confirmed, locally advanced or metastatic NSCLC (adenocarcinoma, bronchoalveolar, squamous cell, large cell, or mixed carcinoma) that is not amendable to surgical treatment and patient has have failed 1 or 2 different lines of chemotherapy.
* Measureable disease and evidence of progression on the previous therapy. Progression may be clinical or radiological.
* ECOG performance status of 0 or 1.
* Life expectancy of at least 3 months.
* Hemoglobin ≥ 10 g/dL.
* Absolute neutrophil count (ANC) ≥ 1500 cells/µL without growth factor support.
* Platelet count ≥ 100,000 cells/µL without support.
* Adequate hepatic and renal function including the following: Total bilirubin < 2 × ULN, AST or ALT ≤ 2.5 × ULN or ≤ 5 × ULN for patients with liver metastasis, PTT within normal limits, INR ≤ 1.5, Serum Creatinine <1.5 ULN
* At least 4 weeks post any radiotherapy or biological therapy; at least 6 weeks post nitrosoureas therapy.
* Full recovery from diagnostic or therapeutic surgery (i.e., complete wound healing) and at least 30 days have elapsed prior to initial dosing.
* Full recovery from the toxic effects of prior therapy (i.e., Common Toxicity Criteria [CTC] Grade 1 or less with the exception of Grade 2 alopecia).
* Women of childbearing potential must have adequate pregnancy test. If postmenopausal, must be ≥ 12 months since last menses.
* Women of childbearing potential and men must agree to use an effective form of contraception during the study and for 60 days after the last dose of study drug.

Exclusion Criteria:

* CNS metastases by radiologic evidence or histology, unless clinically stable (must have been treated by resection or radiation) for at least 4 weeks prior to first dose of study drug. Patients may not be receiving dexamethasone for control of CSF pressure.
* Concurrent therapeutic anticoagulation: PTT less than or equal to 1.5 × ULN or low dose aspirin and low-weight heparin only are allowed.
* More than 2 previous lines of chemotherapy for lung cancer. This includes biologic (immunotherapy) therapy.
* History of previous cerebrovascular accident (CVA) or history transient ischemic attack (TIA) within 6 months of study entry.
* History of prior malignancy not cured by excision. Patients with non-melanoma skin cancer or carcinoma in situ of the cervix are not excluded, but patients with other prior malignancies must have had at least 2-year disease free interval.
* Recent history (within 6 months of screening) of unstable angina, myocardial infarction, or NYHA Class III or IV congestive heart failure
* History of cardiac arrhythmia requiring medical or electrical therapy.
* QTc > 450 msec for males and > 470 msec for females.
* Any major surgery within 30 days or minor surgery within 10 days of study entry, or patient not recovered from surgery.
* History of organ or bone marrow transplant.
* Known active and/or uncontrolled infection, including HIV and are not stable on antiretroviral therapy.
* Any investigational therapy within 28 days of study entry.
* Pregnant or nursing.
* Anyone who in the judgment of the investigator cannot comply with the protocol, provide truly informed consent, or is likely to live < 90 days
* Severe or significant allergy to any chemotherapy or premedication.
* Clinically evident ascites (e.g., abdominal distention, bulging and/or fluid wave) or Grade 3 peripheral edema.
* Any prior cancer treatment with a topoisomerase I inhibitor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2011-06; Primary Completion 2013-02 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: NewLink Genetics, Study Chair — NewLink Genetics Inc
Locations (25):
- Russia (17):
  - State Medical Institution Republican Oncology Center, Saransk, Respublika Mordoviya
  - State Medical Institution Republic Clinical Oncological Center under the Healthcare Ministry of Tatarstan Republic, Kazan', Tatarstan Republic
  - Arkhangelsk Regional Clinical Oncology Center, Arkhangelsk
  - State Healthcare Institution: Bryansk Regional Oncology Center, Bryansk
  - Chelyabinsk Regional Clinical Oncology Center, Chelyabinsk
  - Kursk Regional Oncology Center, Kursk
  - Institution of the Russian Academy of Medical Sciences Russian Oncological Research Center, Moscow
  - Non-Government Medical Institution: Central Clinical Hospital #2, Moscow
  - State Healthcare Institution of Nizhny Novgorod Regiona Nizhny Novgorod Oncology Center, Nizhny Novgorod
  - City Clinical Hospital #1, Novosibirsk
  - State Medical Institution: Pyatigorsk Oncological Center, Pyatigorsk
  - St. Petersburg Medical University, Saint Petersburg
  - City Clinical Oncology Center, Saint Petersburg
  - Stavropol Regional Clinical Oncology Center, Stavropol
  - Tambov Regional Oncology Center, Tambov
  - Primorsky Regional Oncology Center, Vladivostok
  - Regional Clinical Oncology Center, Yaroslavl
- Ukraine (8):
  - Dnipropetrovsk State Medical Academy, Dnipropetrovsk
  - Public Treatment and Prophylaxis Institution; Donetsk Regional Antitumor Center, Donetsk
  - Ivano-Frankovsk State Medical University; Oncology Department Clinical Facility, Ivano-Frankivsk
  - Kharkiv State Public Healthcare Institution: Kharkiv Regional Clinical Oncology Center, Kharkiv
  - Khmelnytskyi Regional Oncology Center, Khmelnytsky
  - Kyiv City Oncology Hospital, Kyiv
  - Sumy Regional Clinical Oncology Center, Sumy
  - Zakarpattia Regional Clinical Oncology Center, Uzhhorod

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted from 04 Jul 2011 to 07 Oct 2014. A total of 24 medical clinics participated in the study.
Groups:
- CRLX101 + BSC (Best Supportive Care): 15 mg/m2 CRLX101 infused IV over 60 minutes every other week + Standard therapy consisting of best supportive care (BSC), including at least blood and platelet transfusions, therapeutic radiation, and bone marrow support (granulocyte colony-stimulating factor [G-CSF]) as required.
- BSC (Best Supportive Care) Alone: Standard therapy consisting of best supportive care (BSC), including at least blood and platelet transfusions, therapeutic radiation, and bone marrow support (granulocyte colony-stimulating factor [G-CSF]) as required.
Period: Overall Study
Arm/Group | CRLX101 + BSC (Best Supportive Care) | BSC (Best Supportive Care) Alone
Started | 100 | 57
Completed | 91 (subjects in ITT with reported date of death, alive with progression, or alive without progression) | 43 (subjects in ITT with reported date of death, alive with progression, or alive without progression)
Not Completed | 9 | 14
Not completed — Withdrawal by Subject | 7 | 11
Not completed — Physician Decision | 1 | 1
Not completed — Adverse Event | 1 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intention-to-treat (ITT) and Patient Safety Population (PSP), includes all CRLX101 + BSC subjects who received at least 1 dose of study treatment and all randomized BSC alone subjects who attended at least 1 study visit.
Groups:
- Total: Total of all reporting groups
Arm/Group | CRLX101 + BSC (Best Supportive Care) | BSC (Best Supportive Care) Alone | Total
Number analyzed (Participants) | 97 | 50 | 147
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58 (8.22) | 60.6 (6.42) | 59.4 (7.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 17 | 42
  Male | 72 | 33 | 105
Region of Enrollment [Number; unit: participants]
  Russian Federation | 56 | 29 | 85
  Ukraine | 41 | 21 | 62

OUTCOME MEASURES:

1. Primary Outcome: To Compare Overall Survival of Patients Treated With CRLX101 + BSC to Those Patients Treated With BSC Only
Description: Comparison of survival among patients treated with CRLX101 + best supportive care vs patients treated wiht best supportive care only.
Time Frame: Up to 18 months
Population: Intention-to-treat (ITT) and Patient Safety Population (PSP), includes all CRLX101 + BSC subjects who received at least 1 dose of study treatment and all randomized BSC alone subjects who attended at least 1 study visit. (Confidence interval if insufficient data to estimate NE = 99999.99)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | CRLX101 | Best Supportive Care
Number analyzed (Participants) | 97 | 50
months | 6.3 [4.70 to 8.68] | 11.9 [6.74 to NA] — Insufficient data to estimate

2. Secondary Outcome: Assess Objective Response Rate (ORR) of CRLX101+ BSC Compared to BSC Only
Description: Comparison of objective response rate in subjects treated with CRLX101+BSC versus subjects treated with BSC alone.
Time Frame: 12 months
Population: Intention-To-Treat (ITT)
Measure: Number; unit: Percentage of Participants
Arm/Group | CRLX101 | Best Supportive Care
Number analyzed (Participants) | 97 | 50
Percentage of Participants | 6.2 | 2.0

ADVERSE EVENTS:
Time Frame: First dose to 30 days after the last dose of study drug
Groups:
- CRLX101+BSC: 15 mg/m2 CRLX101 infused IV over 60 minutes every other week + Standard therapy consisting of best supportive care, including at least blood and platelet transfusions, therapeutic radiation, and bone marrow support (granulocyte colony-stimulating factor [G-CSF]) as required.
- Best Supportive Care (BSC) Only: Standard therapy consisting of best supportive care, including at least blood and platelet transfusions, therapeutic radiation, and bone marrow support (granulocyte colony-stimulating factor [G-CSF]) as required.
Arm/Group | CRLX101+BSC | Best Supportive Care (BSC) Only
Serious Adverse Events (participants affected / at risk) | 12/97 | 5/50
Other Adverse Events (participants affected / at risk) | 76/97 | 39/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CRLX101+BSC (N=97) | Best Supportive Care (BSC) Only (N=50)
atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
cardiopulmonary failure (Cardiac disorders) | 1 (1) | 2 (2)
dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
anaphylatic reaction (Immune system disorders) | 0 (0) | 1 (1)
bronchitis (Infections and infestations) | 2 (2) | 0 (0)
lung abscess (Infections and infestations) | 0 (0) | 1 (1)
pyothorax (Infections and infestations) | 1 (1) | 0 (0)
liver function test (Investigations) | 1 (1) | 0 (0)
psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0)
hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
esophagobronchial fistula (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
superior vena cava syndrome (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CRLX101+BSC (N=97) | Best Supportive Care (BSC) Only (N=50)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 17 (19) | 14 (14)
cough (Respiratory, thoracic and mediastinal disorders) | 14 (14) | 10 (11)
hemoptysis (Respiratory, thoracic and mediastinal disorders) | 7 (10) | 9 (10)
asthenia (General disorders) | 12 (12) | 9 (9)
fatigue (General disorders) | 10 (13) | 4 (4)
chest pain (General disorders) | 8 (8) | 8 (8)
pyrexia (General disorders) | 5 (8) | 5 (9)
pain (General disorders) | 3 (3) | 1 (1)
edema peripheral (General disorders) | 3 (3) | 0 (0)
anemia (Blood and lymphatic system disorders) | 25 (46) | 11 (12)
thrombocytopenia (Blood and lymphatic system disorders) | 5 (18) | 0 (0)
neutropenia (Blood and lymphatic system disorders) | 4 (12) | 0 (0)
leukopenia (Blood and lymphatic system disorders) | 3 (4) | 0 (0)
alanine aminotransferase increased (Investigations) | 8 (11) | 3 (8)
aspartate aminotransferase increased (Investigations) | 8 (14) | 1 (4)
blood creatinine increased (Investigations) | 5 (22) | 1 (1)
blood alkaline phosphatase increased (Investigations) | 3 (3) | 2 (2)
blood glucose increased (Investigations) | 0 (0) | 2 (2)
Eastern Cooperative Oncology Group performance status worsened (Investigations) | 0 (0) | 2 (2)
cystitis (Renal and urinary disorders) | 10 (13) | 2 (3)
hematuria (Renal and urinary disorders) | 7 (9) | 1 (4)
leukocyturia (Renal and urinary disorders) | 5 (8) | 3 (5)
proteinuria (Renal and urinary disorders) | 2 (4) | 2 (2)
nausea (Gastrointestinal disorders) | 11 (19) | 1 (1)
vomiting (Gastrointestinal disorders) | 3 (3) | 1 (1)
diarrhea (Gastrointestinal disorders) | 3 (3) | 0 (0)
bone pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 0 (0)
pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (5) | 0 (0)
back pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 1 (1)
neck pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
pneumonia (Infections and infestations) | 4 (5) | 0 (0)
respiratory tract infection (Infections and infestations) | 2 (2) | 3 (3)
sinus tachycardia (Cardiac disorders) | 0 (0) | 2 (2)
decreased appetitie (Metabolism and nutrition disorders) | 4 (5) | 2 (2)
hyperglycemia (Metabolism and nutrition disorders) | 3 (5) | 2 (2)
headache (Nervous system disorders) | 2 (2) | 3 (3)
dizziness (Nervous system disorders) | 1 (2) | 3 (3)
superior vena cava syndrome (Vascular disorders) | 3 (3) | 0 (0)
hypertension (Vascular disorders) | 3 (4) | 1 (1)
hyperbilirubinemia (Hepatobiliary disorders) | 3 (3) | 2 (5)
alopecia (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) — progression of disease

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigator interested in participating in writing the manuscript should contact the Sponsor. The Investigsator shall not make any Study-related publication or other disclosure without the Sponsor's prior written approval, which may be withheld or granted by the Sponsor, in its sole discretion.